CLINICAL TRIAL: NCT01853137
Title: A Prospective Controlled Evaluation of Class II Division 1 Malocclusions Treated With Fixed Lingual Mandibular Growth Modificator (FLMGM)
Brief Title: Fixed Lingual Mandibular Growth Modificator
Acronym: FLMGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSAMA-18-2-2013
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Class II Division 1 Malocclusion; Retrognathic Mandible
Keywords: Class II division 1 malocclusion; Dentofacial orthopedics; Fixed Lingual Mandibular Growth Modificator (FLMGM)
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLMGM Treatment Group (Experimental)
  Interventions: Device: Fixed Lingual Mandibular Growth Modificator (FLMGM)
- Untreated Class II Control Group (No Intervention)

INTERVENTIONS:
Device: Fixed Lingual Mandibular Growth Modificator (FLMGM) — Novel Class II functional appliance, a fixed version of double-plate appliance
  Other Names: Fixed Lingual Mandibular Growth Modification Appliance (FLMGMA)
  Arms: FLMGM Treatment Group

SUMMARY:
The current trial was designed to investigate the possible initial net skeletal and dental effects of treatment with FLMGM by a comparative evaluation of treated and untreated Cl II/1 malocclusion subjects. The null hypothesis stated that there were no significant differences in dentofacial changes between FLMGM group and control group.

DETAILED DESCRIPTION:
The study was prospective controlled clinical trial conducted at the department of Orthodontics, between May/2009 and June/2011. The protocol of study was approved by the council of scientific research and postgraduate studies.

The original study sample included 43 patients (25 treated, 18 untreated). Of the 43 patients initially enrolled, 38 completed this trial and comprised the final sample, and 5 (4 treated, 1 untreated) were excluded . All patients and parents gave prior informed consent to their inclusion in the investigation.

Patients of both groups were followed on a parallel basis during a period of 8 months and included in the trial regardless of achievement of a Class I incisor relationship. All patient of treatment group (n=21) were treated with FLMGM, and treatment was continued beyond this time point if the Class II malocclusion was not fully corrected and clinical objectives were not achieved. On the other hand, no orthodontic treatment was performed during that duration for the subjects of control group (n=17), and most of control subjects were offered suitable treatment at a later date.

For each patient, a direct digital lateral cephalogram was taken pre- and post- treatment/observation using PAX 400 (VATECH CO., Korea) with the same settings. Cephalograms were digitized on screen and analyzed in a blind manner by the same orthodontist using a cephalometric software (Viewbox, 3.1.1.13, Kifissia). . All linear measurements were reduced to life size (enlargement: 7.54%).

Pretreatment equivalence, changes occurring during the examination period in each group and comparison of changes observed in both groups were tested for significance with t-tests using SPSS . P values of less than 0.05 were considered statistically significant. To assess the method error, twenty cephalograms were randomly picked from both groups and redigitized and analyzed by the same orthodontist after 1 month, and the method error was calculated by Dahlberg's formula.

ELIGIBILITY:
Inclusion Criteria:

Before treatment, each patient fulfilled the following criteria:

1. Cl II/1 malocclusion with an overjet greater than 4 mm.
2. Mild to moderate Class II Skeletal pattern (A-N-B > 4°) with retrognathic mandible (S-N-B < 76°).
3. Growth potential. Fishman skeletal maturation indicator (SMI) method28 was used to assess the hand-wrist radiographs, and only patients in the peak of the pubertal growth spurt, which occurs on average between SMIs 4 to 7,29 at the beginning of the treatment/observation period were invited.

Exclusion Criteria:

-

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osama H Alali, PhD, Principal Investigator — Senior Lecturer, Department of Orthodontics, School of Dentistry, University of Aleppo, Syria
Locations (1):
- Department of Orthodontics, School of Dentistry, University of Damascus, Damascus, Syria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited from those referred to the department of Orthodontics at the University of Damascus between May 2009 and June 2011.
Groups:
- FLMGM Treatment Group: Fixed Lingual Mandibular Growth Modificator (FLMGM) : Novel Class II functional appliance, a fixed version of double-plate appliance
Period: Overall Study
Arm/Group | FLMGM Treatment Group | Untreated Class II Control Group
Started | 25 | 18
Completed | 21 | 17
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Population: Using Bland formula (1995)
Groups:
- Total: Total of all reporting groups
Arm/Group | FLMGM Treatment Group | Untreated Class II Control Group | Total
Number analyzed (Participants) | 25 | 18 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 18 | 43
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (0.9) | 12.5 (2.1) | 13.0 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  Syrian Arab Republic | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Total Mandibular Length (Co-Gn)
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Untreated Class II Control Group: This is a group of patients classified as Class II patients but they are not treated during the observation period of this study
Arm/Group | FLMGM Treatment Group | Untreated Class II Control Group
Number analyzed (Participants) | 21 | 17
mm | 3.51 (1.37) | 1.18 (1.13)

2. Secondary Outcome: Overjet Reduction
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FLMGM Treatment Group | Untreated Class II Control Group
Number analyzed (Participants) | 21 | 17
mm | -3.32 (2.86) | 0.74 (0.94)

ADVERSE EVENTS:
Arm/Group | FLMGM Treatment Group | Untreated Class II Control Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/17
Other Adverse Events (participants affected / at risk) | 0/21 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes